CLINICAL TRIAL: NCT03527238
Title: Optimizing Immunosuppression Drug Dosing Via Phenotypic Precision Medicine
Acronym: PPM - Pro
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB201800053 -N -A; 1R21DK116140-01 (NIH)
Record Dates: First submitted 2018-05-04; First posted 2018-05-17 (Actual); Results first posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Liver Transplant; Kidney Transplant
Keywords: Phenotypic Precision Medicine (PPM); Tacrolimus; Calcineurin Inhibitors
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Standard of Care Tacrolimus Drug Dosing
  Interventions: Drug: Tacrolimus
- Phenotypic Precision Medicine (PPM) (Experimental): PPM-based Computation Assisted Drug Dosing
  Interventions: Other: PPM-based Computation Assisted Drug Dosing; Drug: Tacrolimus

INTERVENTIONS:
Other: PPM-based Computation Assisted Drug Dosing — Tacrolimus dosing based on application of PPM.
  Other Names: Computation based dosing
  Arms: Phenotypic Precision Medicine (PPM)
Drug: Tacrolimus — Dosing of calcineurin inhibitor, tacrolimus

SUMMARY:
Clinical trial applying Phenotypic Precision Medicine (PPM) to tacrolimus dosing in liver and/or kidney transplant recipients to show improvement in maintaining drug trough levels within the target range.

DETAILED DESCRIPTION:
The introduction of calcineurin inhibitors like tacrolimus has greatly reduced the incidence of acute rejection, improving graft and patient survival after transplantation. However, tacrolimus, one of the most widely used immunosuppressants and a mainstay of solid organ transplantation, has a narrow therapeutic index and wide pharmacokinetic variability. As such, there is a clear need for precision medicine to address post-transplant immunosuppression.

The study team has developed a powerful platform [Phenotypic Precision Medicine (PPM)] that utilizes patient-specific clinical data which represents each patient's response to drug treatment. This platform can efficiently prescribe precise and optimized drug doses despite the frequent changes to patient treatment regimens following transplantation. This potentially can have a profound effect on drug metabolism.

The aim of this project is to use PPM to uncover valuable and previously unknown information pertaining to patient dose requirements and correlate them with patient clinical and other contextual information. This study is also expected to reveal vital patient subpopulation information; and any future discovery of quantitative biomarkers as measures of immunosuppression will serve as a gateway towards even more effective personalized and relevant drug dosing.

ELIGIBILITY:
Inclusion Criteria:

* adults undergoing liver and/or kidney transplantation

Exclusion Criteria:

* transplant patients with contraindications to tacrolimus

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Zarrinpar, MD PhD, Principal Investigator — University of Florida
Locations (3):
- United States (2):
  - UCLA, Los Angeles, California
  - UF Health at the University of Florida, Gainesville, Florida
- National University of Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Khong J, Lee M, Warren C, Kim UB, Duarte S, Andreoni KA, Shrestha S, Johnson MW, Battula NR, McKimmy DM, Beduschi T, Lee JH, Li DM, Ho CM, Zarrinpar A. Tacrolimus dosing in liver transplant recipients using phenotypic personalized medicine: A phase 2 randomized clinical trial. Nat Commun. 2025 May 16;16(1):4558. doi: 10.1038/s41467-025-59739-6. PMID 40379675

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | Phenotypic Precision Medicine (PPM)
Started | 31 | 31
Completed | 29 | 27
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Phenotypic Precision Medicine (PPM) | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 25 | 51
  >=65 years | 5 | 6 | 11
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [42 to 61] | 58 [50 to 63] | 57.5 [49.25 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 17 | 18 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 29 | 27 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 29 | 30 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Tacrolimus Target Trough Level Maintenance
Description: Percentage of Days Far (> 2 ng/mL) Out of Range of Tacrolimus Target Trough Level
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Standard of Care | Phenotypic Precision Medicine (PPM)
Number analyzed (Participants) | 29 | 27
percentage of days | 38.4 (27.4) | 24.2 (19.1)

ADVERSE EVENTS:
Time Frame: 30 days after discharge
Arm/Group | Standard of Care | Phenotypic Precision Medicine (PPM)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 6/31 | 6/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=31) | Phenotypic Precision Medicine (PPM) (N=31)
Rejection (Immune system disorders) | 6 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT03527238/Prot_SAP_ICF_001.pdf